CLINICAL TRIAL: NCT01062867
Title: First Administration to Man Of Org 25435 a New Intravenous Anesthetic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Veeda Clinical Research (Industry); Organon Teknika (Unknown)
Responsible Party: Prof J Robert Sneyd, University of Plymouth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 12.4.104
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-01

CONDITIONS: Anaesthesia
Keywords: Anaesthetic
MeSH Terms: interventions — 2-(N-bis(2-methoxyethyl)amino)butyric acid,2',6'-dimethoxyphenyl ester hydrobromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ORG25435 (Experimental): Infusion of intravenous anaesthetic agent to induce anaesthesia
  Interventions: Drug: ORG25435

INTERVENTIONS:
Drug: ORG25435 — Intended doses: 0.25, 0.5, 1.0, 2.0, 3.0, 4.0, 5.0 and 6.0 mg/kg by intravenous infusion over 1 min Up to 25mg/kg by infusion over 30min
  Other Names: ORG 25435

SUMMARY:
Title: First administration to man of Org 25435, a new intravenous anaesthetic.

Protocol: 12.4.104

Clinical Phase: Phase I

Study Site:

Phase I Clinical Trials Unit Ltd Old Convent of Notre Dame 119 Looseleigh Lane Plymouth PL6 5HH United Kingdom

Objectives: To assess the safety, tolerability, preliminary pharmacokinetics and efficacy of Org 25435 as an intravenous anaesthetic.

Study Design: Sequential study of an intravenous anaesthetic in young healthy males, at up to eight dose levels.

Study Drug: Org 25435, a water soluble intravenous anaesthetic.

Subjects: Up to 47 healthy male volunteers, aged 18-40 years.

Evaluations: Tolerability, adverse events, EEG effects, cardiovascular effects, electrocardiogram (ECG), excitatory phenomena, respiratory effects, laboratory safety blood analyses, pharmacodynamic and pharmacokinetic measurements.

DETAILED DESCRIPTION:
Synopsis Trial Number 12.4.104 Trial Title First administration to man of Org 25435 a new intravenous anesthetic Trial Center Phase 1 Clinical Trials Unit Limited, 119 Looseleigh Lane, Derriford, Plymouth PL6 5HH Publication Studied Period The first subject was screened on 04/01/2000 and the final subject completed the follow up on 24/03/2000.

Phase of Development Phase I (First into Man) Objectives To assess the safety, tolerability and efficacy of Org 25435 as an intravenous anesthetic and to obtain preliminary pharmacodynamic and pharmacokinetic details of Org 25435.

Methodology Sequential rising dose study of an intravenous anesthetic in young healthy males, at up to eight dose levels.

Number of Subjects 19 healthy male volunteers were included into the dose escalation part of the study and an additional 7 volunteers participated in the Target Controlled Infusion (TCI) part of the study.

Diagnosis and Main Criteria for Inclusion Inclusion criteria:

Good physical and mental health: absence of a clinically relevant medical history; Clinically acceptable hematology and clinical chemistry results; Hemoglobin > 13.5 g/dl; Normal ECG; Diastolic blood pressure 60 to 90 mmHg inclusive; Normal cardiac morphology demonstrated by echocardiography; Satisfactory cardiovascular response to exercise, measured by the Bruce Protocol, subjects must have completed Bruce stage 5; Aged 18 to 35 years inclusive; Body mass index (BMI) 19 to 27 inclusive, weight 65 to 100 kg inclusive; Negative hepatitis screen; Non-smoker for at least 6 months; Previous experience of general anesthesia with no problems reported; Willingness to give written informed consent; Ability to communicate well with the Investigators.

Investigational Product Dose Mode of Administration Batch Number 1 vial 200mg Org 25435 / 10ml solvent for reconstitution Intended doses: 0.25, 0.5, 1.0, 2.0, 3.0, 4.0, 5.0 and 6.0 mg/kg Intravenous 9J521 Duration of Treatment

Dose Escalation phase:

Each study treatment consisted of an intravenous infusion of Org 25435, given by Infusion pump over exactly 1 minute.

Target Controlled Infusion phase:

Each study treatment consisted of an intravenous infusion of Org25435 given by a computer-controlled infusion over 30 minutes.

Criteria for Evaluation Tolerability, adverse events, EEG effects, cardiovascular effects, electrocardiogram (ECG), excitatory phenomena, respiratory effects, laboratory safety blood analyses, pharmacodynamic and pharmacokinetic measurements. Efficacy Induction phenomena; time of cessation of speech, eye closure, loss of eyelash reflex, eyes open on command, limb movement on command and syringe drop. Other Induction phenomena; pain on injection, sign of histamine release, excitatory phenomena, respiratory depression, apnea. Recovery phenomena; nausea / vomiting, delirium, shivering, disturbed psychomotor function, eye opening on command, spontaneous respiration, adequate respiration, move limbs on command, increased saliva production.

Statistical Methods Formal statistical methods are not appropriate in this small pilot investigative study where group sizes comprise 5 or less subjects. All data collected is presented and summarized according to investigation type (Dose Escalation or TCI).

ELIGIBILITY:
Inclusion Criteria:

* Good physical and mental health:
* Absence of a clinically relevant medical history
* Clinically acceptable hematology and clinical chemistry results
* Hemoglobin > 13.5 g/dl
* Normal ECG
* Diastolic blood pressure 60 to 90 mmHg inclusive
* Normal cardiac morphology demonstrated by echocardiography
* Satisfactory cardiovascular response to exercise, measured by the Bruce Protocol, subjects must have completed Bruce stage 5
* Aged 18 to 35 years inclusive
* Body mass index (BMI) 19 to 27 inclusive, weight 65 to 100 kg inclusive
* Negative hepatitis screen
* Non-smoker for at least 6 months
* Previous experience of general anesthesia with no problems reported -
* Willingness to give written informed consent
* Ability to communicate well with the Investigators.

Exclusion Criteria:

* Females
* History or evidence of clinically significant cardiovascular, respiratory, endocrine, renal, hepatic, neurological or psychiatric disease.
* History of or familial presence of malignant hyperthermia.
* Presence of any condition likely to affect the normal kinetics of the study drug.
* Requirement for prescribed medication.
* Use of concomitant medication in the 5 days prior to dosing.
* General anaesthesia within the previous 3 months.
* History of clinically significant allergy or hypersensitivity to any drug.
* History of clinically significant head injury.
* History of febrile convulsion.
* Known history of human immunodeficiency virus (HIV) infection.
* Use of investigational drug within previous three months.
* Previous administration of an investigational intravenous anaesthetic drug.
* Previous administration of Org 25435 within this study.
* History of alcohol / drug abuse.
* Average consumption of more than 20 units of alcohol a week.
* Subjects who smoke or who have smoked within the past 6 months.
* Inability to communicate with the Investigators for any reason.
* Donation of blood within one month of the study, or the intention to donate blood within one month following the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2000-01; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
induction of anaesthesia (loss of consciousness) | At time of drug administration. Recorded in minutes and seconds from the commencement of infusion.

SECONDARY OUTCOMES:
recovery from anaesthesia (obey verbal commands) | At time of drug administration. Recorded as min and sec from end of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sneyd, MD, Study Chair — University of Plymouth
Locations (2):
- United Kingdom (2):
  - Phase 1 Clinical Trials, Plymouth, Devon
  - Phase 1 Clinical Trials Ltd, Plymouth